CLINICAL TRIAL: NCT00685256
Title: Parent Communication Study II - Randomized Controlled Trial of Decision Support vs. Education for Parent Communication of BRCA 1/2 Cancer Genetic Test Results to Children
Brief Title: Standard Genetic Counseling With or Without a Decision Guide in Improving Communication Between Mothers Undergoing BRCA1/2 Testing and Their Minor-Age Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CDR0000592726; R01HG002686 (NIH); P30CA051008 (NIH); GUMC-2007-444
Record Dates: First submitted 2008-05-24; First posted 2008-05-28 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-02

CONDITIONS: Breast Cancer; Hereditary Breast/Ovarian Cancer (brca1, brca2)
Keywords: breast cancer; hereditary breast/ovarian cancer (BRCA1, BRCA2)
MeSH Terms: conditions — Breast Neoplasms; Hereditary Breast and Ovarian Cancer Syndrome | interventions — Counseling; Early Intervention, Educational; Psychiatric Rehabilitation; Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: counseling intervention — subjects and parents will receive genetic counseling
Other: educational intervention — subjects and parents will receive education re: genetic testing
Other: survey administration — surveys will be administered to subjects and parents
Behavioral: psychosocial assessment and care — psychosocial assessment and counseling will be provided
Behavioral: supportive care — parents and children will be provided with supportive care

SUMMARY:
RATIONALE: A study that evaluates the support of a decision guide used together with genetic counseling may improve communication between mothers undergoing BRCA1/2 testing and their minor-age children.

PURPOSE: This randomized phase III trial is studying standard genetic counseling given together with a decision guide to see how well it works compared with genetic counseling alone in improving communication between mothers undergoing BRCA1/2 testing and their minor-age children.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the efficacy of a decision support intervention delivered in conjunction with standard genetic counseling compared to standard genetic counseling alone in improving communication between mothers undergoing BRCA1/2 testing and their minor-age children.

Secondary

* To understand the mechanisms by which decision support impacts on decision outcomes.
* To identify mothers who are most and least likely to benefit from decision support.
* To explore the potential impact of decision support on disclosure and parent-child psychosocial well-being.

OUTLINE: This is a multicenter study. Mothers are stratified according to their child's age (< 13 vs ≥ 13 years old), child's gender (female vs male), and trial site. Mothers are randomized to 1 of 2 arms.

* Arm I (standard genetic counseling with communication aid): Mothers undergo standard pre-test genetic counseling and provide a blood sample for mutation analysis. Mothers also receive a copy of "My Children, My Test Results," a detailed decision guide developed to promote quality and informed decision making and outcomes, and provide support to mothers regardless of whether or not they choose to communicate their BRCA1/2 test results to their children.
* Arm II (standard genetic counseling alone): Mothers undergo standard pre-test genetic counseling and provide a blood sample for mutation analysis. Mothers also receive a copy of "Genetic Testing for Breast and Ovarian Cancer Risk: It's Your Choice" containing information regarding family history of breast and ovarian cancer risks, BRCA1/2 genes, risks and benefits of genetic testing, medical management options for carriers, and considerations including family communication.

All mothers complete extensive family history assessments during their baseline interviews and disclose if they have been diagnosed with cancer, length and type of treatments, and the number of other relatives with a history of cancer. Mothers are assessed at baseline (pre-test genetic counseling), post-genetic counseling after learning test results, and at 1 and 6 months post-genetic counseling by a 30-45 minute multi-item and multi-scale self-report telephone survey. Genetic testing results are also submitted to this study. The frequency (number), intensity (length in minutes), and content of participant-initiated telephone contacts to genetic counselors to assess intervention reactivity; participants' self-reported use of educational guides; and their satisfaction with the intervention will be assessed.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Mothers self-identified as primary caregivers to minor-age children (ages 8-21 years-old)
* Mothers must be undergoing genetic counseling and have provided a blood sample for analysis for BRCA1/2 mutations
* Mothers must have resided in the same home as the child(ren) for the past 6 months and intend to continue to reside with the child(ren) for the next 6 months

PATIENT CHARACTERISTICS:

* At least 21 years old (mothers)
* No serious mental illness (e.g., cognitive and psychotic disorders) or developmental disability that would limit participation or preclude informed consent
* Must be able to adequately understand, speak, and read English
* Must have ready and consistent access to a telephone

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 8 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2008-03; Primary Completion 2013-02 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Self-reported outcomes at 1-and 6-months | 6 months
Decision conflict, as assessed by the Decisional Conflict Scale | 6 months
Parents' decision satisfaction with their communication decision, as assessed by the Satisfaction With Decision Scale | 6 months
Decision quality | 6 months
Disclosure of genetic testing results by parents | 6 months
Child-rearing alliance between parents, as measured by the Parenting Alliance Measure at baseline, after learning test results, and at 1 and 6 months after genetic counseling | 6 months
Parent-child communication, as assessed by the Parent-Adolescent Communication Scale at baseline, after learning test results, and at 1 and 6 months after genetic counseling | 6 months
Family functioning, as assessed by the Family Relationship Index at baseline, after learning test results, and at 1 and 6 months after genetic counseling | 6 months
Children's stress and worry, as assessed by the Child Behavior Checklist at baseline, after learning test results, and at 1 and 6 months after genetic counseling | 6 months
Parents' knowledge and awareness of the advantages and disadvantages of disclosing maternal BRCA1/2 test results to their children | 6 months
Parents' preferences and values regarding family communication of genetic test results | 6 months
Decision self-efficacy, as assessed by the Decision Self-Efficacy Scale | 6 months
Cognitive appraisals | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Tercyak, PhD, Principal Investigator — Lombardi Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Dana-Farber/Harvard Cancer Center at Dana-Farber Cancer Institute, Boston, Massachusetts